CLINICAL TRIAL: NCT00725660
Title: Pre-Eclampsia Prediction By Doppler Screening Of Uterine Arteries And Angiogenic Factors In Second Trimester Of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: DR. Eyal Mazaki, Shaare Zedek Medical Center Jerusalem Israel
Other Study IDs: 0153-08-HMO.CTIL
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Pregnancy; Pre Eclampsia
Keywords: pre eclampsia; doppler; uterine; arteries; angiogenic; factors
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Pregnant women in second trimester that took the routine triple test, and are having an early routine detailed ultrasound examination.

SUMMARY:
BACKGROUND: Pre-eclampsia complicates about 2% of pregnancies. It accounts for at least 50 000 maternal deaths per year worldwide and is the second most common cause of maternal death in the developing world. Also, Pre-eclampsia is the commonest cause of iatrogenic prematurity, It frequently coexists with intrauterine growth restriction (IUGR) and placental abruption, other important causes of adverse prenatal outcome.

There have been many studies investigating whether the disease can be prevented. In order to achieve this, one needs to be able to identify firstly those women that are at highest risk of the disease.

Early studies showed that impedance to flow in the uterine arteries decreases with gestation in normal pregnancies, while in pregnancies with established pre-eclampsia or IUGR the impedance is increased.

These observations led to a number of screening studies in the second trimester, which assessed if it is possible to predict those pregnancies destined to have complications of impaired placentation. These studies showed that women with increased impedance to uterine artery blood flow have an increased risk of developing pre-eclampsia, and detection can be further increased by using angiogenic factors (That are involved in the pathogenesis of Pre- eclampsia and could be useful for early prediction of the disease: VEGF, PIGF, PP13, sFLT1) in combination with uterine arteries Doppler study in the second trimester.

METHODS: In this study we would like to add uterine arteries Doppler to the early routine detailed ultrasound examination (14-16 weeks), in 3000 women in Jerusalem. in addition we would like to check angiogenic factors from the serum blood taken for the routine triple test in these women (16-18 weeks).pregnancy outcome would be collected after labour from the medical centers participating in this research.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in second trimester that took the routine triple test, and are having an early routine detailed ultrasound examination, in Jerusalem, Israel

Exclusion Criteria:

* none

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women in second trimester that took the routine triple test, and are having an early routine detailed ultrasound examination, in Jerusalem, Israel.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2008-09

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel